CLINICAL TRIAL: NCT03880721
Title: By Developing a Radiomics Model to Predict the Prognosis of Patients With Hepatocellular Carcinoma After Microwave Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Prof., Chinese PLA General Hospital
Other Study IDs: 301jrcsk4
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: radiomics; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Good prognosis
  Interventions: Procedure: Microwave abaltion
- Poor prognosis
  Interventions: Procedure: Microwave abaltion
- Recurrence
  Interventions: Procedure: Microwave abaltion
- Not Recurrence
  Interventions: Procedure: Microwave abaltion
- Survival
  Interventions: Procedure: Microwave abaltion
- Death
  Interventions: Procedure: Microwave abaltion

INTERVENTIONS:
Procedure: Microwave abaltion — Use microwave ablation to treat hepatocellular carcinoma

SUMMARY:
Developing a radiomics model to predict the prognosis of patients with hepatocellular carcinoma after microwave ablation to provide advice for their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hepatocellular carcinoma in the department of interventional ultrasound, PLA general hospital, who accept MWA therapy for HCC

Inclusion criteria:

1. Primary hepatocellular
2. No other treatments ware performed before microwave ablation
3. Patient has been clinically diagnosed with HCC definitely, and have a definite operational indication
4. No extrahepatic manifestations and no evidence of vessel invasion and bile duct thrombi

Exclusion Criteria:

* Exclusion criteria:

  1. Non-primary hepatocellular carcinoma or hepatic metastases
  2. Accept other treatment before microwave ablation
  3. Extrahepatic metastasis, vessel invasion or bile duct thrombi

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
AUC value | through study completion, an average of 2 year
  Utilizing area under curve to judge the accurency
Sensitivity | through study completion, an average of 2 year
  diagnosis sensitivity of intelligent ultrasound analysis
Specificity | through study completion, an average of 2 year
  diagnosis specificity of intelligent ultrasound analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided